CLINICAL TRIAL: NCT05198427
Title: Study MOTIF : mTOR Inhibitors: the Lesions Induced by Papillomavirus for Transplant Patients
Brief Title: mTOR Inhibitors: the Lesions Induced by Papillomavirus for Transplant Patients.
Acronym: MOTIF
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1395
Record Dates: First submitted 2022-01-12; First posted 2022-01-20 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Transplantation Organ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: review of medical patient file — The outcome measure is the evolution of HPV related lesions between :
  * favourable evolution including partial or total regression
  * unfavourable evolution including non-evolution or aggravation or recurrence.

SUMMARY:
The injuries induced by Human Papillomavirus (HPV) (anogenital condyloma mainly) are more frequent among transplanted patients due to their immunosuppression. These injuries are benign but they have a negative impact on the patients' quality of life. The initial treatment is topical and then surgical. The injuries can relapse, especially among transplanted patients.

The modification of the immunosuppressant treatment with a switch to mTOR inhibitors (mammalian Target Of Rapamycin) has shown its efficacy in preventing the recurrence of squamous cell carcinomas or treating Kaposi's disease.

By analogy, this therapeutic strategy can be sometimes put forward to transplanted patients with HPV-induced injuries.

The principal objective of this study is to describe the evolution of HPV-induced lesions in solid organ transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (Age ≥ 18 years)
* Transplanted patient (any organ), having developed HPV-induced lesions after transplantation
* Patient followed or having been followed at Edouard Herriot Hospital (HEH)
* Patient having been informed and not having objected to participating in the study

Exclusion Criteria:

* Transplanted patient without HPV-induced lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient transplanted with HPV-induced lesions from the DIVAT (Validated Transplantation Computerized Data) database for patients followed at the hospital Edouard Herriot
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Evolution of HPV related lesions in patient with switch | at inclusion
  At one year of the switch by an inhibitor of mTOR then remotely of the switch (by tacking the last medical encounter) for the patients concerned by the switch.
Evolution of HPV related lesions in patient without switch | at inclusion
  At one year of the first HPV related lesions care then remotely (by tacking the last medical encounter) for the patients without the switch.

CONTACTS AND LOCATIONS:
Overall Officials: Fanny BURON, MD, Principal Investigator — Hôpital Rdouard Herriot
Locations (1):
- Hôpital Edouard Herriot, Lyon, Auvergne-Rhône-Alpes, France